CLINICAL TRIAL: NCT03323047
Title: Perioperative Tonsillectomy Protocol Development for Preoperative Acetaminophen and Intraoperative High Dose Dexamethasone: a Randomized Control Trial
Brief Title: Perioperative Tonsillectomy Protocol Development
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Josee Paradis, Paediatric Otolaryngologist Assistant Professor - Department of Otolaryngology-Head and Neck Surgery, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 109757
Record Dates: First submitted 2017-10-13; First posted 2017-10-26 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Tonsillitis
Keywords: tonsillectomy; acetaminophen; dexamethasone
MeSH Terms: conditions — Tonsillitis | interventions — Acetaminophen; Dexamethasone; dexamethasone 21-phosphate

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, longitudinal, double-blinded trial at a single centre with 3 groups of 20 children each. Group 1 receives acetaminophen (15 mg/kg) 30 min-1 hr pre-operatively and high-dose dexamethasone (0.5 mg/kg, max. 10 mg) immediately after induction of anesthesia. Group 2 receives acetaminophen (15 mg/kg) 30 min- 1 hr pre-operatively and low-dose dexamethasone (0.15 mg/kg, max. 8 mg) immediately after induction of anesthesia. Group 3 receives placebo 1 hr pre-operatively and low dose dexamethasone (0.15 mg/kg, max. 8 mg) immediately after induction of anesthesia. We will recruit a convenience sample of 60 patients aged 3-13 scheduled for tonsillectomy with the principal investigator or co-investigators. The patients will be placed in one of the groups by a computerized randomization table.
Who Masked: Participant
Masking Description: Participants will blinded to the group that they have been allocated to. Blinding will be possible as all patients will be given either acetaminophen or medication without active ingredients (placebo pilll) and dexamethasone will be administered while the participant is asleep. Participants will be debriefed on which group they were assigned to after all study material is returned (i.e., at their post-operative follow-up appointment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Acetaminophen and High-dose dexamethasone: a single dose of oral acetaminophen (15 mg/kg) 1 hr pre-operatively and intravenous administration of high-dose dexamethasone (0.5 mg/kg, max. 10 mg) immediately after induction of anesthesia.
  Interventions: Drug: Acetaminophen; Drug: High-Dose Dexamethasone
- Group 2 (Active Comparator): Acetaminophen and Low-dose Dexamethasone: a single dose of oral acetaminophen (15 mg/kg) 1 hr pre-operatively and intravenous administration of low-dose dexamethasone (0.15 mg/kg, max. 8 mg) immediately after induction of anesthesia
  Interventions: Drug: Acetaminophen; Drug: Low-dose Dexamethasone
- Group 3 (Placebo Comparator): Placebo oral tablet and Low-dose Dexamethasone: an oral placebo given 1 hr pre-operatively and intravenous administration of low dose dexamethasone (0.15 mg/kg, max. 8 mg) immediately after induction of anesthesia.
  Interventions: Drug: Low-dose Dexamethasone; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Acetaminophen — Oral acetaminophen (15 mg/kg) 1 hr pre-operatively
  Other Names: Tylenol
  Arms: Group 1; Group 2
Drug: Low-dose Dexamethasone — Intravenous low-dose dexamethasone (0.15 mg/kg, max. 8 mg) immediately after induction of anesthesia
  Other Names: Dexamethasone sodium phosphate
  Arms: Group 2; Group 3
Drug: Placebo Oral Tablet — Oral placebo 1 hr pre-operatively
  Other Names: Placebo
  Arms: Group 3
Drug: High-Dose Dexamethasone — Intravenous high-dose dexamethasone (0.5 mg/kg, max. 10 mg) immediately after induction of anesthesia
  Other Names: Dexamethasone sodium phosphate
  Arms: Group 1

SUMMARY:
Pediatric patients who are undergoing a tonsillectomy at the Children's hospital will be randomly assigned to one of three drug groups: 1) acetaminophen (Tylenol) administered pre-operatively and a low dose of anti-inflammatory drug (dexamethasone) administered intra-operatively; 2) acetaminophen (Tylenol) administered pre-operatively and a high dose of anti-inflammatory drug (dexamethasone) administered intra-operatively; 3) no acetaminophen (Tylenol) administered pre-operatively, low dose anti-inflammatory (dexamethasone) administered intra-operatively. The present study will evaluate differences in pain management and surgical complications across the three groups of drug regimens. Main study outcomes include: pain medication administration during surgery, use of pain killers at 1-week post-operation, subjective pain scores administered in the post-anesthesia care unit (PACU) and 1 week postoperation, fluid and food intake, and complication rates (i.e. postoperative bleed rate). The hypothesis is that pain will be lowest in the group that received Tylenol and high-dose dexamethasone (Group 2).

DETAILED DESCRIPTION:
This study will be conducted as a prospective, randomized, longitudinal, double-blinded trial at a single ambulatory surgery centre with 3 groups of 20 children. Group 1 will receive oral acetaminophen (15 mg/kg) 1 hour pre-operatively and high-dose intravenous dexamethasone (0.5 mg/kg, max. dose 10 mg) immediately after induction of anesthesia. Group 2 will receive oral acetaminophen elixir (15 mg/kg) 1 hour pre-operatively and low-dose intravenous dexamethasone (0.15 mg/kg, maximum of 8 mg) immediately after induction of anesthesia. Group 3 will receive an oral placebo 1 hour pre-operatively and low dose intravenous dexamethasone (0.15 mg/kg, maximum of 8 mg) immediately after induction of anesthesia. Dose of dexamethasone is a potential confounder if patients in the low-dose dexamethasone groups weigh enough to obtain the maximum dose (8 mg). We expect this occurrence to be rare, as dexamethasone will be dosed for ideal bodyweight, but subgroup analysis by actual dose received will be performed to compare the two dosing regimens (0.15mg/kg and 0.5 mg/kg).

In addition to these medications, patients will receive the standard peri-operative care at our centre, which consists of intra- operative ondansetron at the discretion of the anesthesiologist, and standing orders for acetaminophen (15 mg/kg) and ibuprofen (10 mg/kg) around the clock. Patients older than five years also receive morphine elixir (0.1 mg/kg rounded down to the nearest 0.5 mg) p.r.n (when necessary) at the discretion of the nurse. Thus, patients of all three groups will receive adequate post-operative symptom control. The Pediatric Otolaryngologist (Dr. Josee Paradis, Dr. Julie Strychowsky, or Dr. Murad Husein) who is the patient's physician and will be performing the tonsillectomy, will initially approach the participant and substitute decision maker (SDM) to describe the study. If the patient and SDM agree to consider the study, the study will be described in more detail and study consent/assent will be obtained by a research assistant or a physician (who is not the primary physician). We will recruit a convenience sample of 60 patients aged 3-13 years scheduled for tonsillectomy to be performed by the principal investigator or co-investigators (J.P., M.H. or J.S.). For children aged 3 to 6 years, SDM informed consent will be obtained; for children aged 7 to 12 years, SDM written consent and child assent will be requested; for children 13 years of age, written consent will be obtained from a SDM and from the child. The patients will be randomized to one of the three treatment groups by a computerized randomization table. Data from the tonsillectomy procedure, including whether analgesia was needed intraoperatively, and in the post-anesthesia care unit, will be recorded. Self-reported pain intensity will be scored on the Oucher tool, a number and picture scale validated in children age 3-13. A research assistant or nurse will be trained to obtain Oucher reports at the patient's bedside at specific post-operative events, which correspond to time points. The Oucher tool is simple to learn and takes minimal time to administer. The first pain report will be obtained once the patient wakes from anesthesia (15 - 45 min post- operation), then upon transfer to step-down care (1 - 2 hrs hour post-operation), then at 3 hours post-operation, and finally upon discharge (or at 5 hours post-operation, if the patient is not anticipated to be discharged by this time). Many of the details surrounding the operation will be gathered in post-hoc review of the patient's chart by the research assistant. If the patient is transferred from the PACU to the day surgery unit (i.e. discharge is anticipated before the end of the day), the information from the entire stay in the day surgery will be collected. If the patient is admitted to the floor (i.e. staying overnight in the hospital for observation), information will be collected from the first 4 hours after admission. The information gathered from the chart will include complications of surgery, whether or not the patient had post-operative bleeding requiring a change in management, and also whether or not the patient had post-operative bleeding that required an operating room procedure. Time to first oral fluid intake, as well as amount of oral intake (measured in quantity of popsicles) in the post-anesthesia care unit and total oral intake before discharge will also be gathered from the patient's chart, as well as the time to first administration of morphine, the dose of morphine required, and the frequency of post-operative vomiting until time of discharge. For home pain management, all patients are advised to take acetominophen (15mg/kg) every 6 hours as needed, alternating with ibuprofen (10mg/kg) every 6 hours as needed. At discharge (average 5 hours post-operation), parents/guardians will be provided with a package including the Pediatric Quality of Life Inventory with questions about oral intake and activity, as well as a space to record any incidents of vomiting, the Oucher tool to evaluate the patient's pain severity, and a medication log to keep track of the pain medication (over the counter or prescribed) that the patient has taken. Parents/guardians will be given a measured cup to record quantity of oral fluid intake for the day. Parents will be asked to fill out the first questionnaire at discharge (average 5 hours post-operation) time point, and they will be encouraged to raise any questions or concerns they have about how to complete the questionnaires. Subsequently, these instruments will be completed by parents/guardians (relationship to patient will be noted on each form and they will be encouraged to have the same parent/guardian complete the form each time) on post-operative days 1, 2, 3, 4, 5, 6, and 7 before bedtime. The research assistant will contact parents/guardians and patients by telephone on the first postoperative day to follow-up with any questions or concerns about the survey. On the last weekday before the patient's follow-up appointment, a reminder call will be made to ask the parent/guardian to bring their completed questionnaire to the appointment. On the 14th post-operative day patients will attend a follow-up visit where they will be assessed and their completed forms will be collected. If the patient had any emergency department visits related to the procedure, the research assistant will consult the hospital database to obtain information about the emergency department visit, including date, chief complaint, and management.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients
* aged 3-13 years
* Level I or level II on the American Society of Anesthesiologists (ASA) physical status classification system (as determined by the anesthesiologist)
* obstructive sleep apnea or recurrent throat infections
* undergoing elective tonsillectomy with or without adenoidectomy
* Parents who agree to complete documentation and follow up at 14 days post-operation.

Exclusion Criteria:

* Patients Level III or greater on the American Society of Anesthesiologists (ASA) physical status classification system (as determined by the anesthesiologist)
* Patients with chronic conditions that would limit our ability to develop the study according to objectives, such as neurodevelopmental conditions preventing patients from understanding the Oucher tool
* Hepatic or renal disease
* cardiac disease
* active infection
* diabetes mellitus
* sickle cell disease
* known coagulation disorders
* pre- operative treatment with anti-emetics, steroids, or analgesics
* Acetaminophen allergy or already receiving acetaminophen within 24 h of surgery
* Complicating health factors precluding the use of opioids or acetaminophen
* any other factors which would interfere with pain assessment and management
* Patients weighing more than 30 kg that would exceed maximum dexamethasone dose
* Patients who live without a home telephone
* patient living without parental supervision.

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Oucher pain score | awakening from anesthesia (0.5 hours post- operation)
  pain intensity on the Oucher pain tool, which includes ratings by face scale and a number scale (0-10).

SECONDARY OUTCOMES:
Analgesia use | during operation
  Whether or not intraoperative analgesia was required
time to first oral fluid intake | during patient's stay in PACU (on average 5 hours)
  amount of time that elapses before patient has a fluid intake
time to first request for morphine | during patient's stay in PACU (on average 5 hours)
  the time that elapses before patient requests morphine (if applicable)
dose of morphine required | from end of operation to 7 days post-operation
  if morphine administered, frequency, dosage and total amount of morphine patient took post-operatively
vomiting | From end of operation to 7 days post-operation
  Number of times patient vomited after surgery
Pediatric Quality of Life Inventory | Upon discharge (on average 5 hours post-operation), and 1 day, 2 days, 3 days, 4 days, 5 days, 6 days, 7 days post-operation
  Validated post-tonsillectomy Quality of life questionnaire with Likert-scale questions regarding common post-operative symptoms
Medication log | discharge (on average 5 hours post-operation) to 7 days post-operation
  Record of pain medications (over the counter and prescription) patient as taken post-discharge from hospital
Oucher pain score | transfer to step-down care (1 hour post-operation), 3 hours post-operation, 5 hours post-operation, upon discharge, as well as 1 day, 2 days, 3 days, 4 days, 5 days, 6 days, 7 days post-operation
  pain intensity on the Oucher pain tool, which includes ratings by face scale and a number scale (0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Josee Paradis, MD, Principal Investigator — LHSC
Locations (1):
- Children's Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No